CLINICAL TRIAL: NCT05333835
Title: A 26-week, Randomized, Open-label, 3-arm Parallel, Treat-to-target Study Comparing the Efficacy and Safety of HR17031 Injection to INS068 Injection and to SHR20004 Injection in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin With or Without One Other Oral Anti-diabetic Drug
Brief Title: A Trial Comparing the Efficacy and Safety of HR17031 Injection to INS068 Injection and to SHR20004 Injection in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR17031-201
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: HR17031 injection compared with Ins068 injection and SHR20004 injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HR17031 injection (Experimental)
  Interventions: Drug: HR17031 injection
- INS068 injection (Active Comparator)
  Interventions: Drug: INS068 injection
- SHR20004 injection (Active Comparator)
  Interventions: Drug: SHR20004 injection

INTERVENTIONS:
Drug: HR17031 injection — HR17031 injection
  Arms: HR17031 injection
Drug: INS068 injection — INS068 injection
  Arms: INS068 injection
Drug: SHR20004 injection — SHR20004 injection
  Arms: SHR20004 injection

SUMMARY:
The aim of this trial is to compare the efficacy and safety of HR17031 versus INS068 and SHR20004 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-70 age years, both inclusive;
2. BMI is 20.0 to 40.0 kg/m2, both inclusive;
3. Type 2 diabetes mellitus diagnosed for at least 3 months before the screening visit;
4. HbA1c 7.5-11.0% (both inclusive) by local laboratory analysis;
5. At screening:

1) Treatment with metformin alone on a stable dose (≥1500 mg or at the maximum tolerated dose [MTD, ≥1000 mg]) for ≥3 months, or 2) Treatment with metformin at the above dose level combined with a second OAD (AGI, SU, TZD, glinides, DPP-4i or SGLT2i) on a stable dose (≥half of the max approved dose according to local label, or at the MTD) for ≥3 months.

Exclusion Criteria:

1. Use of systemic glucocorticoids within 3 months prior to the screening;
2. Use of weight loss drugs within 3 months prior to the screening.
3. Treatment with insulin within 1 year prior to screening (except for short-term or treatment for gestational diabetes);
4. Laboratory findings at the screening visit:

   * Amylase and/or lipase >3 x upper limit of normal (ULN);
   * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 x ULN;
   * Moderate (3b) or severe renal failure or renal insufficiency or according to local contraindications for metformin;
   * Urinary albumin creatinine ratio (UACR) ≥300 mg/g;
   * Total bilirubin >2.0 x ULN;
   * Calcitonin ≥50 ng/L;
5. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)；
6. Cardiac disorder defined as: congestive heart failure (NYHA class III-IV), diagnosis of unstable angina pectoris, cerebral stroke and/or myocardial infarction within the last 6 months prior to screening and/or planned coronary, carotid or peripheral artery revascularization procedures;
7. Severe uncontrolled treated or untreated hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg);
8. Proliferative retinopathy, maculopathy, painful diabetic neuropathy, diabetic foot ulcer or intermittent claudication requiring acute treatment;
9. History of pancreatitis (acute or chronic);
10. Pregnancy, breast-feeding, intention of becoming pregnant during the trial; or women of childbearing potential (WOCBP) or male subject not using adequate contraceptive measures；

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in HbA1c at Week 26 | at Week 26

SECONDARY OUTCOMES:
Mean Change From Baseline in fasting plasma glucose (FPG) at Week 26 | at Week 26
Mean Change From Baseline in Body Weight at Week 26 | at Week 26
Proportion of subjects reaching HbA1c targets (<7.0%; ≤6.5%) at Week 26 | at Week 26
Mean Actual Daily Insulin Dose at Week 26 | at Week 26
Number of Hypoglycaemic Episodes at Week 26 | at Week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided